CLINICAL TRIAL: NCT00393484
Title: A Phase IV Study of the Antiviral Activity and Safety of Entecavir Versus Lamivudine in Adults With Chronic Hepatitis B Infection Who Are Negative for Hepatitis B e Antigen in Korea
Brief Title: A Study in Korea of Entecavir Versus Lamivudine in Adults With Chronic Hepatitis B Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AI463-105
Record Dates: First submitted 2006-10-26; First posted 2006-10-27 (Estimated); Results first posted 2010-11-18 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-11

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir; Lamivudine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm A (Experimental): Entecavir + Lamivudine placebo (0-96 weeks)
  Entecavir (96-240 weeks)
  Interventions: Drug: Entecavir; Drug: Lamivudine Placebo
- Arm B (Active Comparator): Lamivudine + Entecavir placebo (0-96 weeks)
  Lamivudine (96-240 weeks)
  Interventions: Drug: Lamivudine; Drug: Entecavir Placebo

INTERVENTIONS:
Drug: Entecavir — Tablets, Oral, 0.5 mg, once daily (0-96 weeks) and (96-240 weeks)
  Other Names: Baraclude; BMS-200475
  Arms: Arm A
Drug: Lamivudine Placebo — Capsules, Oral, 0 mg, once daily (0-96 weeks)
  Arms: Arm A
Drug: Lamivudine — Capsules, Oral, 100 mg, once daily (0-96 weeks)
  Tablets, Oral, 100 mg, once daily (96-240 weeks)
  Arms: Arm B
Drug: Entecavir Placebo — Tablets, Oral, 0 mg, once daily (0-96 weeks)
  Arms: Arm B

SUMMARY:
Entecavir, 0.5 mg daily, will have clinical efficacy (assessed as an undetectable hepatitis B DNA, <300 copies/mL, by Roche Comprehensive Bio-Analytical System Amplicor polymerase chain reaction assay) that is comparable (noninferior) and potentially superior to lamivudine, 100 mg once daily, in adults with hepatitis B e antigen-negative chronic hepatitis B virus infection.

ELIGIBILITY:
Inclusion Criteria:

* Nucleoside and nucleotide-naive subjects with chronic HBV infection
* Hepatitis B Surface antigen(HBsAg)-positive ≥6 months
* Detectable HBsAg
* HBV DNA ≥ 105 copies/mL by PCR
* ALT 1.3 to 10 x the ULN
* HBeAg negative, anti-hepatitis B Virus E antigen antibody (anti-HBeAb) positive status

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2007-02; Primary Completion 2009-01 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (8):
- South Korea (8):
  - Local Institution, Bucheon-si
  - Local Institution, Busan
  - Local Institution, Chuncheon
  - Local Institution, Daegu
  - Local Institution, Daejeon
  - Local Institution, Guri-si
  - Local Institution, Jeonju
  - Local Institution, Seoul

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 122 participants were enrolled in this study; 2 did not receive treatment.
Groups:
- Entecavir, 0.5 mg + Placebo: Participants received entecavir, 0.5 mg, once daily, with lamivudine placebo tablets, once daily, administered orally through Week 96 (double-blind period). Then, participants received entecavir, 0.5 mg, once daiy, administered orally for Weeks 96-240 (open-label period).
- Lamivudine, 100 mg + Placebo: Participants received lamivudine, 100 mg, once daily, with entecavir placebo tablets, once daily, administered orally, through Week 96 (double-blind period). Then, participants received lamivudine, 0.5 mg, once daiy, administered orally for Weeks 96-240 (open-label period).
Period: Double-blind Period (Day 1 to Week 96)
Arm/Group | Entecavir, 0.5 mg + Placebo | Lamivudine, 100 mg + Placebo
Started | 56 (Number treated) | 64 (Number treated)
Participants Excluded From Analysis | 1 | 1
Completed | 54 | 52
Not Completed | 2 | 12
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — No longer met inclusion criteria | 0 | 3
Not completed — Lack of Efficacy | 0 | 6
Not completed — Lost to Follow-up | 0 | 2
Period: Open-label Period (Weeks 96 to 240)
Arm/Group | Entecavir, 0.5 mg + Placebo | Lamivudine, 100 mg + Placebo
Started | 48 | 44
Withdrew Consent | 6 (Did not participate in open-label period) | 6 (Did not participate in open-label period)
Lack of Efficacy | 0 (Did not participate in open-label period) | 2 (Did not participate in open-label period)
Completed | 40 | 21
Not Completed | 8 | 23
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 1 | 2
Not completed — Noncompliance | 2 | 2
Not completed — Lack of Efficacy | 0 | 18

BASELINE CHARACTERISTICS:
Population: All participants who received study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | Entecavir, 0.5 mg + Placebo | Lamivudine, 100 mg + Placebo | Total
Number analyzed (Participants) | 56 | 64 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.73 (11.93) | 48.98 (7.84) | 47.46 (10.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 16 | 25
  Male | 47 | 48 | 95
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 56 | 64 | 120
Prior interferon treatment status [Number; unit: Participants]
  No | 54 | 64 | 118
  Yes | 2 | 0 | 2
Hepatitis B virus DNA by polymerase chain reaction [Mean (Standard Deviation); unit: log10 copies/mL] | 6.06 (0.78) | 5.79 (0.90) | 5.91 (0.86)
Alanine aminotransferase [Mean (Standard Deviation); unit: U/L] | 110.46 (81.97) | 93.94 (58.46) | 101.65 (70.59)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved a Virologic Response at Week 24
Description: Virologic response=Hepatitis B virus DNA <300 copies/mL by polymerase chain reaction assay.
Time Frame: At Week 24
Population: Randomized participants who received at least 1 dose of study drug
Measure: Number; unit: Percentage of participants
Arm/Group | Entecavir, 0.5 mg + Placebo | Lamivudine, 100 mg + Placebo
Number analyzed (Participants) | 56 | 64
Percentage of participants | 92.86 | 67.19
Statistical Analysis 1: Comparison: Entecavir, 0.5 mg + Placebo vs Lamivudine, 100 mg + Placebo; A sample size of 60 per group provides 80% power for testing superiority of entecavir compared to lamivudine, assuming a response rate of 62% for lamivudine and 83% for entecavir; Test type: Non-Inferiority or Equivalence — The difference in proportion along with its standard error and 90% confidence interval was computed. If the lower limit of the confidence interval (CI) was great than -10%, noninferiority was established. Provided that noninferiority was established, a test for superiority was planned to check that the lower limit of the 90% CI was greater than zero; p = 0.0006, Chi-squared — There was no adjustment for the prior test of noninferiority because the test for superiority could succeed only if noninferiority was first established; Difference in proportion = 25.67, 90% CI 2-sided [14.48 to 36.86]

2. Secondary Outcome: Number of Participants With Hepatitis B Virus (HBV) DNA <10^3, <10^4, or < 10^5 Copies/mL by Polymerase Chain Reaction (PCR) Assy at Weeks 24, 48, and 96
Description: The number and percentage of participants achieving the following endpoints will be tabulated at each visit through Week 240 by treatment group: HBV DNA <300 copies/mL by PCR assay; HBV DNA <10^3, <10^4, or < 10^5 copies/mL by PCR assay. Treatment comparisons will be assessed using the same method as the primary endpoint.
Time Frame: At Weeks 24, 48, and 96
Population: Randomized participants who received at least 1 dose of study drug
Measure: Number; unit: Participants
Arm/Group | Entecavir, 0.5 mg + Placebo | Lamivudine, 100 mg + Placebo
Number analyzed (Participants) | 56 | 64
Participants
  Week 24: HBV DNA <10^3 | 54 | 46
  Week 24: HBV DNA <10^4 | 54 | 53
  Week 24: HBV DNA <10^5 | 54 | 59
  Week 48: HBV DNA <10^3 | 54 | 45
  Week 48: HBV DNA <10^4 | 55 | 50
  Week 48: HBV DNA <10^5 | 55 | 52
  Week 96: HBV DNA <10^3 | 53 | 38
  Week 96: HBV DNA <10^4 | 53 | 42
  Week 96: HBV DNA <10^5 | 53 | 45
Statistical Analysis 1: Comparison: Entecavir, 0.5 mg + Placebo vs Lamivudine, 100 mg + Placebo; HBV DNA <10^3 copies/mL at 24 Weeks; Test type: Superiority or Other; p = 0.0003, Chi-squared — Treatment comparisons were assessed using the same method used in the primary endpoint; Difference = 24.55, 90% CI 2-sided [14.45 to 34.66]
Statistical Analysis 2: Comparison: Entecavir, 0.5 mg + Placebo vs Lamivudine, 100 mg + Placebo; HBV DNA <10^4 copies/mL at 24 Weeks; Test type: Superiority or Other; p = 0.0167, Chi-squared — Treatment comparisons were assessed using the same method as the primary endpoint; Difference = 13.62, 90% CI 2-sided [4.85 to 22.38]
Statistical Analysis 3: Comparison: Entecavir, 0.5 mg + Placebo vs Lamivudine, 100 mg + Placebo; HBV DNA <10^5 at 24 Weeks; Test type: Superiority or Other; p = 0.4467, Chi-squared; Mean Difference (Final Values) = 4.24, 90% CI 2-sided [-2.62 to 11.10]
Statistical Analysis 4: Comparison: Entecavir, 0.5 mg + Placebo vs Lamivudine, 100 mg + Placebo; HBV DNA <10^3 copies/mL at 48 Weeks; Test type: Superiority or Other; p = 0.0002, Chi-squared; Difference = 26.12, 90% CI 2-sided [15.87 to 36.36]
Statistical Analysis 5: Comparison: Entecavir, 0.5 mg + Placebo vs Lamivudine, 100 mg + Placebo; HBV DNA <10^4 copies/mL at 48 Weeks; Test type: Superiority or Other; p = 0.0009, Chi-squared; Difference = 20.09, 90% CI 2-sided [11.10 to 29.07]
Statistical Analysis 6: Comparison: Entecavir, 0.5 mg + Placebo vs Lamivudine, 100 mg + Placebo; HBV DNA <10^5 at 48 Weeks; Test type: Superiority or Other; p = 0.0029, Chi-squared; Difference = 16.96, 90% CI 2-sided [8.43 to 25.50]
Statistical Analysis 7: Comparison: Entecavir, 0.5 mg + Placebo vs Lamivudine, 100 mg + Placebo; HBV DNA <10^3 copies/mL at 96 Weeks; Test type: Superiority or Other; p < 0.0001, Chi-squared; Difference = 35.27, 90% CI 2-sided [24.02 to 46.51]
Statistical Analysis 8: Comparison: Entecavir, 0.5 mg + Placebo vs Lamivudine, 100 mg + Placebo; HBV DNA <10^4 copies/mL at 96 Weeks; Test type: Superiority or Other; p < 0.0001, Chi-squared; Difference = 29.02, 90% CI 2-sided [18.07 to 39.97]
Statistical Analysis 9: Comparison: Entecavir, 0.5 mg + Placebo vs Lamivudine, 100 mg + Placebo; HBV DNA <10^5 copies/mL at 96 Weeks; Test type: Superiority or Other; p = 0.0006, Chi-squared; Difference = 24.33, 90% CI 2-sided [13.71 to 34.95]

3. Secondary Outcome: Mean Log10 Reduction From Baseline in Hepatitis B Virus (HBV) DNA at Weeks 24, 48, 96, 144, 192, and 240
Description: Mean log10 reduction from Baseline in HBV DNA virus by the Roche Comprehensive Bio-Analytical System Amplicor polymerase chain reaction (PCR) assay at Week 24. The extent of the decrease was estimated by comparing HBV DNA levels of all participants in each group with a linear regression model with covariates of treatment and baseline HBV DNA by PCR assay.
Time Frame: At Weeks 24, 48, 96, 144, 192, and 240
Population: Randomized participants who received at least 1 dose of study drug
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Groups:
- Lamivudine, 100 mg+ Placebo: Participants received lamivudine, 100 mg, once daily, with entecavir placebo tablets, once daily, administered orally, through Week 96 (double-blind period). Then, participants received lamivudine, 0.5 mg, once daiy, administered orally for Weeks 96-240 (open-label period).
Arm/Group | Entecavir, 0.5 mg + Placebo | Lamivudine, 100 mg+ Placebo
Number analyzed (Participants) | 56 | 64
log10 copies/mL
  At 24 Weeks | 3.58 (0.60) | 2.95 (0.69)
  At 48 Weeks | 3.56 (0.53) | 2.65 (0.61)
  At 96 Weeks | 3.59 (0.52) | 2.42 (0.60)
  At 144 Weeks | -3.60 (0.60) | -2.74 (0.70)
  At 192 Weeks | -3.60 (0.63) | -2.75 (0.73)
  At 240 Weeks | -3.53 (0.85) | -2.69 (0.98)
Statistical Analysis 1: Comparison: Entecavir, 0.5 mg + Placebo vs Lamivudine, 100 mg+ Placebo; Changes from baseline were based on patients with measurements at both Baseline and Week 24; Test type: Superiority or Other; p < 0.0001, unpaired t-test — Treatment comparisons were based on 2-sided t-test for treatment difference (entecavir: lamivudine) estimated from the linear regression model with covariates of treatment and baseline hepatitis B DNA by PCR
Statistical Analysis 2: Comparison: Entecavir, 0.5 mg + Placebo vs Lamivudine, 100 mg+ Placebo; Changes from Baseline were based on patients with measurements at both Baseline and at Week 48; Test type: Superiority or Other; p < 0.0001, unpaired t-test — Treatment comparisons were based on 2-sided t-test for treatment difference (entecavir: lamivudine) estimated from the linear regression model with covariants of treatment and Baseline hepatitis B DNA by PCR
Statistical Analysis 3: Comparison: Entecavir, 0.5 mg + Placebo vs Lamivudine, 100 mg+ Placebo; Changes from Baseline were based on patients with measurements at both Baseline and at 96 Weeks; Test type: Superiority or Other; p < 0.0001, unpaired t-test — [p-value comment as in outcome 3, analysis 2]
Statistical Analysis 4: Comparison: Entecavir, 0.5 mg + Placebo vs Lamivudine, 100 mg+ Placebo; Changes from Baseline were based on patients with measurements at both Baseline and at Week 144; Test type: Superiority or Other; p < 0.0001, unpaired t-test — [p-value comment as in outcome 3, analysis 2]
Statistical Analysis 5: Comparison: Entecavir, 0.5 mg + Placebo vs Lamivudine, 100 mg+ Placebo; Changes from Baseline were based on patients with measurements at both Baseline and at Week 192; Test type: Superiority or Other; p < 0.0001, unpaired t-test — [p-value comment as in outcome 3, analysis 2]
Statistical Analysis 6: Comparison: Entecavir, 0.5 mg + Placebo vs Lamivudine, 100 mg+ Placebo; Changes from Baseline were based on patients with measurements at both Baseline and at Week 240; Test type: Superiority or Other; p < 0.0001, unpaired t-test — [p-value comment as in outcome 3, analysis 2]

4. Secondary Outcome: Mean Laboratory Test Values for Alanine Aminotransferase (ALT) at Week 24
Description: Mean ALT values from baseline by laboratory test. .
Time Frame: At Week 24
Population: Randomized participants who received at least 1 dose of study drug
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Entecavir, 0.5 mg + Placebo | Lamivudine, 100 mg + Placebo
Number analyzed (Participants) | 56 | 64
U/L | 31.5 (14.04) | 43.26 (32.08)

5. Secondary Outcome: Number of Participants With Normalization of Serum Alanine Aminotransferase (ALT) Levels at Weeks 24, 48, and 96
Description: Normalization of serum ALT= ≤*institutional upper limit of normal.
Time Frame: At Weeks 24, 48, and 96
Population: Randomized participants who received at least 1 dose of study drug
Measure: Number; unit: Participants
Arm/Group | Entecavir, 0.5 mg + Placebo | Lamivudine, 100 mg + Placebo
Number analyzed (Participants) | 56 | 64
Participants
  At 24 Weeks | 43 | 37
  At 48 Weeks | 48 | 38
  At 96 Weeks | 49 | 33
Statistical Analysis 1: Comparison: Entecavir, 0.5 mg + Placebo vs Lamivudine, 100 mg + Placebo; Test type: Superiority or Other; p = 0.0278, Chi-squared; Difference = 18.97, 90% CI 2-sided [5.22 to 32.73] — At 24 Weeks
Statistical Analysis 2: Comparison: Entecavir, 0.5 mg + Placebo vs Lamivudine, 100 mg + Placebo; Test type: Superiority or Other; p = 0.0014, Chi-squared; Difference = 26.34, 90% CI 2-sided [13.65 to 39.03] — At 48 Weeks
Statistical Analysis 3: Comparison: Entecavir, 0.5 mg + Placebo vs Lamivudine, 100 mg + Placebo; Test type: Superiority or Other; p < 0.0001, Chi-squared; Difference = 35.94, 90% CI 2-sided [23.35 to 48.52] — At 96 Weeks

6. Secondary Outcome: Number of Participants With Death as Outcome, Serious Adverse Events (SAEs), Discontinuations Due to Adverse Events (AEs), Most Common AEs, and Grade 3/4 AEs at Week 24
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Most common AEs=AEs affecting ≥3 participants. Grade 3 (Severe)/Grade 4 (Very Severe)AEs per World Health Organization (WHO) criteria.Serious adverse events/deaths reported for enrolled patients regardless of treatment status.
Time Frame: Start of dosing (Day 1) until end of treatment (Week 24) + 5 days and to end of 24-week follow-up period
Population: Treated cohort: includes participants who are randomized and received at least 1 dose of study drug (ETV or LVD).
Measure: Number; unit: Participants
Arm/Group | Entecavir, 0.5 mg + Placebo | Lamivudine, 100 mg + Placebo
Number analyzed (Participants) | 56 | 64
Participants
  Deaths | 0 | 0
  SAEs | 0 | 3
  Discontinuations Due to AEs | 0 | 1
  Any AEs | 14 | 23
  Most common AEs: Upper Respiratory Infection | 3 | 7
  Most common AEs: Nasopharyngitis | 1 | 4
  Most common AEs: Urticaria | 0 | 3
  WHO Grade 3/4 AEs | 0 | 0

7. Secondary Outcome: Number of Participants With Elevations in Alanine Transaminase (ALT) and Aspartate Aminoaminase (AST) Levels, Elevations in ALT and AST Levels,Simultaneous Elevations in ALT and Total Bilirubin Levels, and ALT Flares at Week 24
Description: ALT flares=ALT>2*Baseline and 10*upper limit of normal. Serious adverse events/deaths reported for enrolled patients regardless of treatment status.
Time Frame: Start of dosing (Day 1) until end of treatment (24 weeks) + 5 days and to end of 24-week follow-up period
Population: Randomized participants who received at least 1 dose of study drug
Measure: Number; unit: Participants
Arm/Group | Entecavir, 0.5 mg + Placebo | Lamivudine, 100 mg + Placebo
Number analyzed (Participants) | 56 | 64
Participants
  ALT elevations >2*Baseline (BL) | 0 | 1
  AST elevations >2*BL | 0 | 1
  ALT elevations >3*BL & AST elevations >2*BL | 0 | 1
  Simultaneous ALT & Total bilirubin elevation | 0 | 0
  ALT flares | 0 | 0

8. Secondary Outcome: Number of Participants With Grade 3 or 4 Abnormalities in Laboratory Test Results by World Health Organization (WHO) Criteria at Week 24
Description: ULN=upper limit of normal; ALT=alanine transaminase. WHO criteria: Grade 3=Severe (inability to carry out usual activity); Grade 4=Very severe (debilitating or significantly incapacitating patient despite symptomatic treatment).
Time Frame: Start of dosing (Day 1) until end of treatment (Week 24) + 5 days and to the end of the 24-week follow-up period
Population: Randomized participants who received at least 1 dose of study drug
Measure: Number; unit: Participants
Arm/Group | Entecavir, 0.5 mg + Placebo | Lamivudine, 100 mg + Placebo
Number analyzed (Participants) | 56 | 64
Participants
  Gr 4 Prothrombin time (>3*ULN) | 1 | 0
  Gr 3 Glucose (251-500 mg/dL) | 1 | 2
  Gr 3 ALT (5.1-10*ULN) | 0 | 1
  Gr 3 Lipase (2.0-5.0*ULN) | 0 | 1

9. Secondary Outcome: Number of Participants With Clinically or Statistically Significant Changes in Vital Sign Measurements at Week 24
Description: Vital signs assessed included blood pressure, heart rate, body temperature, and respiration rate.
Time Frame: Start of dosing (Day 1) until end of treatment (Week 24) + 5 days and to end of 24-week follow-up period
Population: Randomized participants who received at least 1 dose of study drug
Measure: Number; unit: Participants
Arm/Group | Entecavir, 0.5 mg + Placebo | Lamivudine, 100 mg + Placebo
Number analyzed (Participants) | 56 | 64
Participants | 0 | 0

10. Secondary Outcome: Number of Participants With Virologic Rebound at Week 24
Description: Virologic rebound was defined as a confirmed ≥1 log10 increase in hepatitis B virus (HBV) DNA from nadir on blinded treatment (as determined by 2 sequential HBV DNA measurements or last on-treatment measurement).
Time Frame: At Week 24
Measure: Number; unit: Participants
Groups:
- Lamivudine, 100 mg: Participants received lamivudine, 100 mg, once daily for up to 240 weeks
Arm/Group | Entecavir, 0.5 mg + Placebo | Lamivudine, 100 mg
Number analyzed (Participants) | 56 | 64
Participants | 0 | 3

11. Secondary Outcome: Percentage of Participants With a Virologic Response as Defined by Undetectable Hepatitis B Virus DNA at Weeks 48, 96, 144, 192, and 240
Description: Undetectable HBV DNA= <300 copies/mL by polymerase chain reaction assay
Time Frame: At Weeks 48, 96, 144, 192, and 240
Population: Randomized participants who received at least 1 dose of study drug
Measure: Number; unit: Percetage of participants
Arm/Group | Entecavir, 0.5 mg + Placebo | Lamivudine, 100 mg + Placebo
Number analyzed (Participants) | 56 | 64
Percetage of participants
  At 48 Weeks | 94.64 | 60.94
  At 96 Weeks | 94.64 | 48.44
  At 144 Weeks | 67.86 | 34.38
  At 192 Weeks | 69.64 | 25.00
  At 240 Weeks | 67.86 | 15.63
Statistical Analysis 1: Comparison: Entecavir, 0.5 mg + Placebo vs Lamivudine, 100 mg + Placebo; Test type: Superiority or Other; p < 0.0001, Chi-squared; Difference = 33.71, 90% CI 2-sided [22.52 to 44.89] — At 48 Weeks
Statistical Analysis 2: Comparison: Entecavir, 0.5 mg + Placebo vs Lamivudine, 100 mg + Placebo; Test type: Superiority or Other; p < 0.0001, Chi-squared; Mean Difference (Final Values) = 46.21, 90% CI 2-sided [34.80 to 57.61] — At 96 Weeks
Statistical Analysis 3: Comparison: Entecavir, 0.5 mg + Placebo vs Lamivudine, 100 mg + Placebo; Test type: Superiority or Other; p = 0.0003, Chi-squared; Difference = 33.48, 90% CI 2-sided [19.31 to 47.65] — At 144 Weeks
Statistical Analysis 4: Comparison: Entecavir, 0.5 mg + Placebo vs Lamivudine, 100 mg + Placebo; Test type: Superiority or Other; p < 0.0001, Chi-squared; Difference = 44.64, 90% CI 2-sided [31.17 to 58.11] — At 192 Weeks
Statistical Analysis 5: Comparison: Entecavir, 0.5 mg + Placebo vs Lamivudine, 100 mg + Placebo; Test type: Superiority or Other; p < 0.0001, Chi-squared; Difference = 52.23, 90% CI 2-sided [39.54 to 64.93] — At 240 Weeks

12. Secondary Outcome: Number of Participants With Viral Rebound and Drug-resistant Hepatitis B Virus (HBV) DNA Mutations at Week 96
Description: Virologic rebound was defined as a confirmed ≥1 log10 increase in HBV DNA from nadir on blinded treatment (as determined by 2 sequential HBV DNA values or last on-treatment measurement).
Time Frame: At 96 weeks
Population: All participants who received study drug and who had samples of measureable HBV DNA values
Measure: Number; unit: Participants
Arm/Group | Entecavir, 0.5 mg + Placebo | Lamivudine, 100 mg + Placebo
Number analyzed (Participants) | 55 | 61
Participants
  Viral rebound | 1 | 26
  Drug-resistant mutations | 0 | 13
Statistical Analysis 1: Comparison: Entecavir, 0.5 mg + Placebo vs Lamivudine, 100 mg + Placebo; Viral rebound at 96 weeks; Test type: Superiority or Other; p < 0.0001, Chi-squared

13. Secondary Outcome: Number of Participants With Death as Outcome, Serious Adverse Events (SAEs), Discontinuations Due to Adverse Events (AEs), Most Common AEs, and Grade 3/4 AEs at Week 240
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization.
Time Frame: Start of dosing (Day 1) until end of treatment (Week 240) + 5 days
Population: Participants who were randomized and received at least 1 dose of study drug
Measure: Number; unit: Participants
Arm/Group | Entecavir, 0.5 mg + Placebo | Lamivudine, 100 mg + Placebo
Number analyzed (Participants) | 56 | 64
Participants
  SAEs | 7 | 17
  Discontinuations due to AEs | 0 | 1
  Any nonserious AEs | 48 | 49
  Nonserious AEs related to study conditions | 1 | 6
  SAEs related to study conditions | 0 | 0

14. Secondary Outcome: Number of Participants With Grade 3 or 4 Abnormalities in Laboratory Test Results by World Health Organization (WHO) Criteria at Week 96
Description: as for outcome 8
Time Frame: Start of dosing (Day 1) until Week 96
Population: Randomized participants who received at least 1 dose of study drug and who were evaluable.
Measure: Number; unit: Participants
Arm/Group | Entecavir, 0.5 mg + Placebo | Lamivudine, 100 mg + Placebo
Number analyzed (Participants) | 55 | 62
Participants
  Platelets | 1 | 1
  Prothrombin time | 1 | 0
  Neutrophils | 0 | 1
  AST | 0 | 3
  ALT | 0 | 6
  Total bilirubiin | 1 | 3
  Creatinine | 2 | 0
  Lipase | 2 | 4
  Potassium | 0 | 1
  Glucose, fasting | 3 | 2

ADVERSE EVENTS:
Time Frame: Start of dosing (Day 1) until end of treatment (Week 240) + 5 days
Groups:
- Entecavir , 0.5 mg + Placebo: Participants received entecavir, 0.5 mg, once daily, with lamivudine placebo tablets, once daily, administered orally through Week 96 (double-blind period). Then, participants received entecavir, 0.5 mg, once daiy, administered orally for Weeks 96-240 (open-label period).
Arm/Group | Entecavir , 0.5 mg + Placebo | Lamivudine, 100 mg + Placebo
Serious Adverse Events (participants affected / at risk) | 7/56 | 17/64
Other Adverse Events (participants affected / at risk) | 28/56 | 29/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Entecavir , 0.5 mg + Placebo (N=56) | Lamivudine, 100 mg + Placebo (N=64)
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Liposarcoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Subdural hemorrhage (Injury, poisoning and procedural complications) | 2 | 0
Blood glucose increased (Investigations) | 1 | 0
Gallbladder polyp (Hepatobiliary disorders) | 1 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 1
Tibia fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pituitary tumor benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Cerebral vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Intervertebral disc herniation (Musculoskeletal and connective tissue disorders) | 0 | 1
Red blood cell count decreased (Investigations) | 0 | 1
Chondrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colonic polyp (Gastrointestinal disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hydrocephalus (Nervous system disorders) | 1 | 0
Optic neuropathy (Eye disorders) | 1 | 0
Subarachnoid hemorrhage (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Entecavir , 0.5 mg + Placebo (N=56) | Lamivudine, 100 mg + Placebo (N=64)
Upper respiratory tract infection (Infections and infestations) | 9 | 12
Nasopharyngitis (Infections and infestations) | 6 | 6
Colonic polyp (Gastrointestinal disorders) | 0 | 3
Fatigue (General disorders) | 5 | 6
Insomnia (Psychiatric disorders) | 2 | 3
Blood glucose increased (Investigations) | 0 | 3
Reflux esophagitis (Gastrointestinal disorders) | 3 | 2
Dermatitis, contact (Skin and subcutaneous tissue disorders) | 1 | 3
Gastritis (Gastrointestinal disorders) | 5 | 2
Hepatic enzyme increased (Investigations) | 0 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Dyspepsia (Gastrointestinal disorders) | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.